CLINICAL TRIAL: NCT05724095
Title: Electrical Acupoint Stimulation Alleviates Hypotension After Spinal Anesthesia in Parturients: a Prospective Randomized Controlled Clinical Trial
Brief Title: Electrical Acupoint Stimulation Reduces Intrathecal Anesthesia Induced Hypotension
Acronym: EARTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhihong LU (Other)
Responsible Party: Sponsor-Investigator, Zhihong LU, Associate professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJH-20230203
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Hypotension During Surgery
Keywords: transcutaneous electrical acupoint stimulation; spinal anesthesia; hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Sham Comparator)
  Interventions: Other: electrodes attached
- low frequency stimulation (Experimental)
  Interventions: Other: low frequency acupoint stimulation; Other: electrodes attached
- high frequency stimulation (Experimental)
  Interventions: Other: high frequency acupoint stimulation; Other: electrodes attached

INTERVENTIONS:
Other: high frequency acupoint stimulation — electrodes are attached to area of acupoints and electrical stimulation at 10/50 Hz is given
  Arms: high frequency stimulation
Other: low frequency acupoint stimulation — electrodes are attached to area of acupoints and electrical stimulation at 2/10 Hz is given
  Arms: low frequency stimulation
Other: electrodes attached — electrodes are attached to area of acupoints

SUMMARY:
The parturients may suffer from hypotension after spinal anesthesia and the incidence could be as high as 70-80% when pharmacological prophylaxis is not used. Acupuncture was reported to treat hypotension both in human and animal studies. Possible mechanisms include modulating cardiovascular and sympathetic system. In this prospective, double-blinded, randomized clinical trial, we tend to investigate the effect of transcutaneous electric acupoint stimulation (TEAS) on hypotension in parturients undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* American Society of Anesthesiologists physical status Ⅰ-Ⅱ
* singleton pregnancy
* full-term gestation (≥38 weeks)

Exclusion Criteria:

* Parturients suffering from preeclampsia
* Parturients with hypertension, diabetes, or cardiac dysfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
incidence of hypotension by 30 minutes after spinal anesthesia | from injection of anesthetics to 30 minutes after injection, in a total of 30 minutes
  Hypotension episodes, defined as reductions in systolic blood pressure exceeding 30% of baseline or <90 mm Hg

SECONDARY OUTCOMES:
lowest systolic blood pressure during 30 minutes after spinal anesthesia | from injection of anesthetics to 30 minutes after injection, in a total of 30 minutes
dose of ephedrine | from injection of anesthetics to 30 minutes after injection, in a total of 30 minutes
  hypotension is treated with ephedrine in increments of 10 mg every 2 minutes
nausea and vomiting score | from injection of anesthetics to 30 minutes after injection, in a total of 30 minutes
  The presence of nausea and vomiting is measured on a 3-point scale of 1, 2, and 3, indicating no nausea and no vomiting, nausea only, and both nausea and vomiting, respectively.
incidence of dizzy | from injection of anesthetics to 30 minutes after injection, in a total of 30 minutes
incidence of apnea | from injection of anesthetics to 30 minutes after injection, in a total of 30 minutes
incidence of chest congestion | from injection of anesthetics to 30 minutes after injection, in a total of 30 minutes
dose of atropine | from injection of anesthetics to 30 minutes after injection, in a total of 30 minutes
  Heart rate lower than 50 beats per minute is treated with 0.5mg of atropine
Apgar score at 1 minute | 1minute after birth
  Apgar score of the neonates at 1minute after birth. The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Fourth military medical university, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arai YC, Kato N, Matsura M, Ito H, Kandatsu N, Kurokawa S, Mizutani M, Shibata Y, Komatsu T. Transcutaneous electrical nerve stimulation at the PC-5 and PC-6 acupoints reduced the severity of hypotension after spinal anaesthesia in patients undergoing Caesarean section. Br J Anaesth. 2008 Jan;100(1):78-81. doi: 10.1093/bja/aem306. Epub 2007 Oct 24. PMID 17959591
- [Result] Adigun TA, Amanor-Boadu SD, Soyannwo OA. Comparison of intravenous ephedrine with phenylephrine for the maintenance of arterial blood pressure during elective caesarean section under spinal anaesthesia. Afr J Med Med Sci. 2010 Mar;39(1):13-20. PMID 20632667
- [Result] Chooi C, Cox JJ, Lumb RS, Middleton P, Chemali M, Emmett RS, Simmons SW, Cyna AM. Techniques for preventing hypotension during spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD002251. doi: 10.1002/14651858.CD002251.pub4. PMID 32619039
- [Derived] Liu X, Gao Z, Jiang Y, Tuo X, He S, Xu F, Lu Z. Comparison of Low-Frequency or High-Frequency Electrical Acupoint Stimulation on Hypotension After Spinal Anesthesia in Parturients: A Prospective Randomized Controlled Clinical Trial. J Integr Complement Med. 2024 Aug;30(8):770-775. doi: 10.1089/jicm.2023.0610. Epub 2024 Mar 28. PMID 38546428